CLINICAL TRIAL: NCT03214861
Title: Carbohydrate Quality and Quantity and Risk of Coronary Heart Disease Among US Women and Men.
Brief Title: Carb Quality and CHD in US Adults
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Kuwait Foundation for the Advancement of Science (Unknown); National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Hala Alessa, Research Fellow, Harvard School of Public Health (HSPH)
Other Study IDs: Carb Quality and CHD NHS HPFS; UM1CA186107 (NIH); UM1CA167552 (NIH); HL34594 (Other Grant/Funding Number: NHLBI); HL35464 (Other Grant/Funding Number: NHLBI); DK58845 (Other Grant/Funding Number: NIDDK); KFAS012016 (Other Grant/Funding Number: Kuwait Foundation for the Advancement of Science)
Record Dates: First submitted 2017-07-10; First posted 2017-07-12 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-07

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nurses Health Study: The Nurses' Health Study (NHS) was initiated in 1976 as a prospective cohort study, where 121,701 female registered nurses between the ages of 30 and 55 years were recruited from 11 US states.
  Interventions: Other: Carbohydrate quality
- Health Professionals Follow-Up Study: The Health Professionals Follow-up Study (HPFS) was initiated in 1986 and recruited 51,529 US men between the ages of 40-75.
  Interventions: Other: Carbohydrate quality

INTERVENTIONS:
Other: Carbohydrate quality — This is an observational study examining the association between carbohydrate quality and coronary heart disease. The investigators used a variety of carbohydrate quality metrics to evaluate carbohydrate quality including carbohydrate, starch, total fiber, cereal fiber, fruit fiber, and vegetable fiber intakes, and the ratios of carbohydrate to total fiber, carbohydrate to cereal fiber, starch to total fiber, and starch to cereal fiber intakes.

SUMMARY:
This is an analysis conducted in the Nurses Health Study and the Health Professional Follow-Up Study, both prospective cohort studies, where the investigators systematically investigated the association between carbohydrate quality using a variety of metrics in relation to coronary heart disease. This was a secondary data analysis of previously collected data in both cohorts.

DETAILED DESCRIPTION:
In this study, the investigators studied the association between carbohydrate quality and coronary heart disease using prospective cohort studies among US adults. Carbohydrate quality was evaluated using a variety of metrics including carbohydrate, starch, total fiber, cereal fiber, fruit fiber, and vegetable fiber intake, as well as the ratios of carbohydrate to total fiber, carbohydrate to cereal fiber, starch to total fiber, and starch to cereal fiber. The Nurses' Health Study (NHS) and the Health Professionals Follow Up Study (HPFS) started in 1984 and 1986, respectively, and were followed-up every 2-4 years thereafter until 2012. Participants include in this study had up to 28y of follow-up. All participants were free of known diabetes mellitus, cancer or cardiovascular disease at baseline. Cox proportional hazards regression models were used to assess the relationship between dietary measures of carbohydrate quality and incident CHD (nonfatal myocardial infarction and fatal CHD).

ELIGIBILITY:
Inclusion Criteria:

* Participants of these two cohorts

Exclusion Criteria:

* Participants with diabetes, coronary heart disease, or cancer at baseline
* Participants with missing exposure information at baseline
* Participants with implausible food frequency questionnaire info (females: kcal < 500 or > 3500; males: kcal < 800 or > 4200)
* Participants who left 10 or more items blank on the food frequency questionnaire

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The analysis was based on two cohorts: one of female registered nurses and the other of male health professionals only.
Study Population: The Nurses' Health Study (NHS) was initiated in 1976 as a prospective cohort study, where 121,701 female registered nurses between the ages of 30 and 55 years were recruited from 11 US states. The Health Professionals Follow-up Study (HPFS) was initiated in 1986 and recruited 51,529 US men between the ages of 40-75. Every two years, participants updated their information on medical history, lifestyle, and incidence of chronic diseases using validated questionnaires. Follow-up rates are at least 90% of potential person-years of follow-up and mortality follow-up is more than 98%.
Sampling Method: Non-Probability Sample
Enrollment: 117885 (Actual)
Dates: Start 1976-06 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Coronary Heart Disease (CHD) | June 1984 - June 2012
  CHD includes both fatal and non-fatal myocardial infarction

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] Huffman MD, Capewell S, Ning H, Shay CM, Ford ES, Lloyd-Jones DM. Cardiovascular health behavior and health factor changes (1988-2008) and projections to 2020: results from the National Health and Nutrition Examination Surveys. Circulation. 2012 May 29;125(21):2595-602. doi: 10.1161/CIRCULATIONAHA.111.070722. Epub 2012 Apr 30. PMID 22547667
- [Background] Yang L, Colditz GA. Prevalence of Overweight and Obesity in the United States, 2007-2012. JAMA Intern Med. 2015 Aug;175(8):1412-3. doi: 10.1001/jamainternmed.2015.2405. No abstract available. PMID 26098405
- [Background] Long-Term Trends in Diagnosed Diabetes. CDC's Division of Diabetes Translation. National Diabetes Surveillance System. October 2011. http://www.cdc.gov/diabetes/statistics
- [Background] Mozumdar A, Liguori G. Persistent increase of prevalence of metabolic syndrome among U.S. adults: NHANES III to NHANES 1999-2006. Diabetes Care. 2011 Jan;34(1):216-9. doi: 10.2337/dc10-0879. Epub 2010 Oct 1. PMID 20889854
- [Background] Stampfer MJ, Hu FB, Manson JE, Rimm EB, Willett WC. Primary prevention of coronary heart disease in women through diet and lifestyle. N Engl J Med. 2000 Jul 6;343(1):16-22. doi: 10.1056/NEJM200007063430103. PMID 10882764
- [Background] Akesson A, Larsson SC, Discacciati A, Wolk A. Low-risk diet and lifestyle habits in the primary prevention of myocardial infarction in men: a population-based prospective cohort study. J Am Coll Cardiol. 2014 Sep 30;64(13):1299-306. doi: 10.1016/j.jacc.2014.06.1190. PMID 25257629
- [Background] U.S. Department of Agriculture and the U.S. Department of Health and Human Services. Nutrition and your health. Dietary guidelines for Americans. 1980.
- [Background] McGuire S. U.S. Department of Agriculture and U.S. Department of Health and Human Services, Dietary Guidelines for Americans, 2010. 7th Edition, Washington, DC: U.S. Government Printing Office, January 2011. Adv Nutr. 2011 May;2(3):293-4. doi: 10.3945/an.111.000430. Epub 2011 Apr 30. No abstract available. PMID 22332062
- [Background] Siri-Tarino PW, Sun Q, Hu FB, Krauss RM. Meta-analysis of prospective cohort studies evaluating the association of saturated fat with cardiovascular disease. Am J Clin Nutr. 2010 Mar;91(3):535-46. doi: 10.3945/ajcn.2009.27725. Epub 2010 Jan 13. PMID 20071648
- [Background] Li Y, Hruby A, Bernstein AM, Ley SH, Wang DD, Chiuve SE, Sampson L, Rexrode KM, Rimm EB, Willett WC, Hu FB. Saturated Fats Compared With Unsaturated Fats and Sources of Carbohydrates in Relation to Risk of Coronary Heart Disease: A Prospective Cohort Study. J Am Coll Cardiol. 2015 Oct 6;66(14):1538-1548. doi: 10.1016/j.jacc.2015.07.055. PMID 26429077
- [Background] Yu D, Shu XO, Li H, Xiang YB, Yang G, Gao YT, Zheng W, Zhang X. Dietary carbohydrates, refined grains, glycemic load, and risk of coronary heart disease in Chinese adults. Am J Epidemiol. 2013 Nov 15;178(10):1542-9. doi: 10.1093/aje/kwt178. Epub 2013 Sep 5. PMID 24008907
- [Background] Rebello SA, Koh H, Chen C, Naidoo N, Odegaard AO, Koh WP, Butler LM, Yuan JM, van Dam RM. Amount, type, and sources of carbohydrates in relation to ischemic heart disease mortality in a Chinese population: a prospective cohort study. Am J Clin Nutr. 2014 Jul;100(1):53-64. doi: 10.3945/ajcn.113.076273. Epub 2014 Apr 30. PMID 24787492
- [Background] Liu S, Willett WC, Stampfer MJ, Hu FB, Franz M, Sampson L, Hennekens CH, Manson JE. A prospective study of dietary glycemic load, carbohydrate intake, and risk of coronary heart disease in US women. Am J Clin Nutr. 2000 Jun;71(6):1455-61. doi: 10.1093/ajcn/71.6.1455. PMID 10837285
- [Background] Yang Q, Zhang Z, Gregg EW, Flanders WD, Merritt R, Hu FB. Added sugar intake and cardiovascular diseases mortality among US adults. JAMA Intern Med. 2014 Apr;174(4):516-24. doi: 10.1001/jamainternmed.2013.13563. PMID 24493081
- [Background] Lloyd-Jones DM, Hong Y, Labarthe D, Mozaffarian D, Appel LJ, Van Horn L, Greenlund K, Daniels S, Nichol G, Tomaselli GF, Arnett DK, Fonarow GC, Ho PM, Lauer MS, Masoudi FA, Robertson RM, Roger V, Schwamm LH, Sorlie P, Yancy CW, Rosamond WD; American Heart Association Strategic Planning Task Force and Statistics Committee. Defining and setting national goals for cardiovascular health promotion and disease reduction: the American Heart Association's strategic Impact Goal through 2020 and beyond. Circulation. 2010 Feb 2;121(4):586-613. doi: 10.1161/CIRCULATIONAHA.109.192703. Epub 2010 Jan 20. PMID 20089546
- [Background] Mozaffarian RS, Lee RM, Kennedy MA, Ludwig DS, Mozaffarian D, Gortmaker SL. Identifying whole grain foods: a comparison of different approaches for selecting more healthful whole grain products. Public Health Nutr. 2013 Dec;16(12):2255-64. doi: 10.1017/S1368980012005447. Epub 2013 Jan 4. PMID 23286205
- [Background] AlEssa HB, Bhupathiraju SN, Malik VS, Wedick NM, Campos H, Rosner B, Willett WC, Hu FB. Carbohydrate quality and quantity and risk of type 2 diabetes in US women. Am J Clin Nutr. 2015 Dec;102(6):1543-53. doi: 10.3945/ajcn.115.116558. Epub 2015 Nov 4. PMID 26537938
- [Background] Hu FB, Stampfer MJ, Rimm E, Ascherio A, Rosner BA, Spiegelman D, Willett WC. Dietary fat and coronary heart disease: a comparison of approaches for adjusting for total energy intake and modeling repeated dietary measurements. Am J Epidemiol. 1999 Mar 15;149(6):531-40. doi: 10.1093/oxfordjournals.aje.a009849. PMID 10084242
- [Background] Willett WC, Sampson L, Stampfer MJ, Rosner B, Bain C, Witschi J, Hennekens CH, Speizer FE. Reproducibility and validity of a semiquantitative food frequency questionnaire. Am J Epidemiol. 1985 Jul;122(1):51-65. doi: 10.1093/oxfordjournals.aje.a114086. PMID 4014201
- [Background] Salvini S, Hunter DJ, Sampson L, Stampfer MJ, Colditz GA, Rosner B, Willett WC. Food-based validation of a dietary questionnaire: the effects of week-to-week variation in food consumption. Int J Epidemiol. 1989 Dec;18(4):858-67. doi: 10.1093/ije/18.4.858. PMID 2621022
- [Background] Rimm EB, Giovannucci EL, Stampfer MJ, Colditz GA, Litin LB, Willett WC. Reproducibility and validity of an expanded self-administered semiquantitative food frequency questionnaire among male health professionals. Am J Epidemiol. 1992 May 15;135(10):1114-26; discussion 1127-36. doi: 10.1093/oxfordjournals.aje.a116211. PMID 1632423
- [Background] Feskanich D, Rimm EB, Giovannucci EL, Colditz GA, Stampfer MJ, Litin LB, Willett WC. Reproducibility and validity of food intake measurements from a semiquantitative food frequency questionnaire. J Am Diet Assoc. 1993 Jul;93(7):790-6. doi: 10.1016/0002-8223(93)91754-e. PMID 8320406
- [Background] Willett WC. Nutritional Epidemiology. New York: Oxford University Press, 1998.
- [Background] Nutrient Data Laboratory (U.S.), Consumer and Food Economics Institute (U.S.), USDA nutrient database for standard reference. Riverdale, MD.: USDA Nutrient Data Laboratory, Agricultural Research Service, 1999:CD-ROMs.
- [Background] Willett WC, Howe GR, Kushi LH. Adjustment for total energy intake in epidemiologic studies. Am J Clin Nutr. 1997 Apr;65(4 Suppl):1220S-1228S; discussion 1229S-1231S. doi: 10.1093/ajcn/65.4.1220S. PMID 9094926
- [Background] Rose GA, Blackburn H. Cardiovascular survey methods. Monogr Ser World Health Organ. 1968;56:1-188. No abstract available. PMID 4972212
- [Background] Jr. FEH. Regression Modeling Strategies: Applications to Linear Models, Logistic Regression, and Survival Analysis. New York, NY.: Springer-Verlag, 2001.
- [Background] McKeown NM, Meigs JB, Liu S, Rogers G, Yoshida M, Saltzman E, Jacques PF. Dietary carbohydrates and cardiovascular disease risk factors in the Framingham offspring cohort. J Am Coll Nutr. 2009 Apr;28(2):150-8. doi: 10.1080/07315724.2009.10719766. PMID 19828900
- [Background] Yang Y, Zhao LG, Wu QJ, Ma X, Xiang YB. Association between dietary fiber and lower risk of all-cause mortality: a meta-analysis of cohort studies. Am J Epidemiol. 2015 Jan 15;181(2):83-91. doi: 10.1093/aje/kwu257. Epub 2014 Dec 31. PMID 25552267
- [Background] Rimm EB, Ascherio A, Giovannucci E, Spiegelman D, Stampfer MJ, Willett WC. Vegetable, fruit, and cereal fiber intake and risk of coronary heart disease among men. JAMA. 1996 Feb 14;275(6):447-51. doi: 10.1001/jama.1996.03530300031036. PMID 8627965
- [Background] Zong G, Gao A, Hu FB, Sun Q. Whole Grain Intake and Mortality From All Causes, Cardiovascular Disease, and Cancer: A Meta-Analysis of Prospective Cohort Studies. Circulation. 2016 Jun 14;133(24):2370-80. doi: 10.1161/CIRCULATIONAHA.115.021101. PMID 27297341
- [Background] Johnsen NF, Frederiksen K, Christensen J, Skeie G, Lund E, Landberg R, Johansson I, Nilsson LM, Halkjaer J, Olsen A, Overvad K, Tjonneland A. Whole-grain products and whole-grain types are associated with lower all-cause and cause-specific mortality in the Scandinavian HELGA cohort. Br J Nutr. 2015 Aug 28;114(4):608-23. doi: 10.1017/S0007114515001701. Epub 2015 Jul 23. PMID 26201847
- [Background] Wu H, Flint AJ, Qi Q, van Dam RM, Sampson LA, Rimm EB, Holmes MD, Willett WC, Hu FB, Sun Q. Association between dietary whole grain intake and risk of mortality: two large prospective studies in US men and women. JAMA Intern Med. 2015 Mar;175(3):373-84. doi: 10.1001/jamainternmed.2014.6283. PMID 25559238
- [Background] Liu S, Stampfer MJ, Hu FB, Giovannucci E, Rimm E, Manson JE, Hennekens CH, Willett WC. Whole-grain consumption and risk of coronary heart disease: results from the Nurses' Health Study. Am J Clin Nutr. 1999 Sep;70(3):412-9. doi: 10.1093/ajcn/70.3.412. PMID 10479204
- [Background] Tang G, Wang D, Long J, Yang F, Si L. Meta-analysis of the association between whole grain intake and coronary heart disease risk. Am J Cardiol. 2015 Mar 1;115(5):625-9. doi: 10.1016/j.amjcard.2014.12.015. Epub 2014 Dec 18. PMID 25727082
- [Background] Barclay AW, Petocz P, McMillan-Price J, Flood VM, Prvan T, Mitchell P, Brand-Miller JC. Glycemic index, glycemic load, and chronic disease risk--a meta-analysis of observational studies. Am J Clin Nutr. 2008 Mar;87(3):627-37. doi: 10.1093/ajcn/87.3.627. PMID 18326601
- [Background] Jenkins DJ, Wolever TM, Leeds AR, Gassull MA, Haisman P, Dilawari J, Goff DV, Metz GL, Alberti KG. Dietary fibres, fibre analogues, and glucose tolerance: importance of viscosity. Br Med J. 1978 May 27;1(6124):1392-4. doi: 10.1136/bmj.1.6124.1392. PMID 647304
- [Background] Howarth NC, Saltzman E, Roberts SB. Dietary fiber and weight regulation. Nutr Rev. 2001 May;59(5):129-39. doi: 10.1111/j.1753-4887.2001.tb07001.x. PMID 11396693
- [Background] Lutsey PL, Jacobs DR Jr, Kori S, Mayer-Davis E, Shea S, Steffen LM, Szklo M, Tracy R. Whole grain intake and its cross-sectional association with obesity, insulin resistance, inflammation, diabetes and subclinical CVD: The MESA Study. Br J Nutr. 2007 Aug;98(2):397-405. doi: 10.1017/S0007114507700715. Epub 2007 Mar 29. PMID 17391554
- [Background] Ferrannini E, Buzzigoli G, Bonadonna R, Giorico MA, Oleggini M, Graziadei L, Pedrinelli R, Brandi L, Bevilacqua S. Insulin resistance in essential hypertension. N Engl J Med. 1987 Aug 6;317(6):350-7. doi: 10.1056/NEJM198708063170605. PMID 3299096
- [Background] Laws A, Reaven GM. Evidence for an independent relationship between insulin resistance and fasting plasma HDL-cholesterol, triglyceride and insulin concentrations. J Intern Med. 1992 Jan;231(1):25-30. doi: 10.1111/j.1365-2796.1992.tb00494.x. PMID 1732395
- [Background] Juhan-Vague I, Alessi MC, Joly P, Thirion X, Vague P, Declerck PJ, Serradimigni A, Collen D. Plasma plasminogen activator inhibitor-1 in angina pectoris. Influence of plasma insulin and acute-phase response. Arteriosclerosis. 1989 May-Jun;9(3):362-7. doi: 10.1161/01.atv.9.3.362. PMID 2470343
- [Derived] AlEssa HB, Cohen R, Malik VS, Adebamowo SN, Rimm EB, Manson JE, Willett WC, Hu FB. Carbohydrate quality and quantity and risk of coronary heart disease among US women and men. Am J Clin Nutr. 2018 Feb 1;107(2):257-267. doi: 10.1093/ajcn/nqx060. PMID 29529162